CLINICAL TRIAL: NCT00987740
Title: A Prospective, Non-Randomized Feasibility Study of the Hemolung Respiratory Assist System in COPD Patients With Acute Respiratory Failure That Are at a 50% Risk of Failing Non Invasive Ventilation (NIV)
Brief Title: Feasibility Study of the Hemolung Respiratory Assist System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alung Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-CA-2000
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Hypercapnic Respiratory Failure, COPD
Keywords: hypercapnic respiratory failure, COPD
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Hemolung Respiratory Assist System (Experimental)
  Interventions: Device: Hemolung Respiratory Assist System

INTERVENTIONS:
Device: Hemolung Respiratory Assist System — Patients meeting the inclusion criteria will be placed on the Hemolung Respiratory Assist System. Patients will be weaned from non-invasive ventilation and then the Hemolung. Hemolung support will be provided for up to 7 days. Follow-up exams will be performed every 15 days until hospital discharge or 30 days from completion of Hemolung therapy, whichever is later.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Hemolung Respiratory Assist System in patients with hypercapnic respiratory failure associated with acute exacerbation of chronic obstructive pulmonary disease (COPD) and a 50% likelihood of failure of noninvasive positive pressure ventilation leading to intubation and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe COPD, as defined by the GOLD criteria
* Acute exacerbation of COPD (sustained worsening of patient's condition necessitating a change in regular medication)
* On non-invasive positive pressure mechanical ventilation > 1hour with either:
* PaCO2 > 55 mmHg with pH < 7.25 OR
* PaCO2 > 55 mmHg with < 5mmHg decrease from baseline and pH < 7.30
* Not severely hypoxemic (PaO2/FiO2 ≥ 200 mmHg on PEEP/CPAP ≤ 5 cmH2O)
* Hemodynamically stable (mean arterial pressure > 65 mmHg without vasopressor support)
* Chronic arrhythmias (e.g., atrial fibrillation) well controlled
* Minimum platelet count of 100,000/mm3
* Minimum red blood cell count of 2.5 mill/μl

Exclusion Criteria:

* Presence of acute, uncontrolled arrhythmia
* Acute ischemic heart disease
* Presence of bleeding diathesis
* Significant abnormality or weakness/paralysis of respiratory muscles due to a know muscular dystrophy or neurologic disorder
* Recent (< 7 days) prolonged (>24 hrs) use of muscle paralyzing agents
* Cerebrovascular accident, intracranial bleed, head injury or other neurologic disorder likely to affect ventilation
* Coma from any cause, or decreased consciousness
* Hypersensitivity to heparin or previous heparin induced thrombocytopenia
* Recent (< 6 months) major chest abdominal trauma or surgery
* Presence of septic shock
* Presence of a significant pneumothorax or bronchopleural fistula
* History of uncontrolled major psychiatric disorder
* Pregnant women
* Known to have AIDS or to have symptomatic HIV
* Received chemotherapy or radiation within the previous 90 days
* Received an organ transplant other than corneal transplants
* Received or currently receiving immunosuppressive therapy, excluding corticosteroids within the last 3 months
* Presence of severe renal or liver failures
* Known vascular abnormality with could complicate or prevent successful insertion of the vascular access catheter in the right femoral vein
* Presence of another catheter in the right femoral vein that cannot be moved
* Presence of an inferior vena cava filter

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of serious adverse events while on Hemolung therapy and up to 30 days after cessation of therapy and decannulation. | 30 days
Percentage of patients requiring Mechanical Ventilation | 7 days

SECONDARY OUTCOMES:
Improvement in patient self assessment of dyspnea using visual analog scale pre- to post-Hemolung therapy. | 7 days
Change in Minute Volume (VE) pre- to end-Hemolung therapy | 7 days
Number of days in the ICU | 30 days
Number of days in the hospital | 30 days
Number of days alive and off mechanical ventilation for > 48 hours through the end of Day 30 following completion of Hemolung therapy | 30 days
Percentage of patients requiring sedation, and hours of sedation | 30 days
Number of days on Non-Invasive Positive Pressure Ventilation (NIPPV) | 30 days
For patients requiring Mechanical Ventilation, number of days on Mechanical Ventilation | 30 days
Duration of weaning time from NIPPV | 7 days
Duration of weaning time from Hemolung therapy | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: RK Mani, MD, Principal Investigator — Artemis Health Institute
Locations (1):
- Artemis Health Institute, Gurgaon, Haryana, India

REFERENCES:
- [Derived] Burki NK, Mani RK, Herth FJF, Schmidt W, Teschler H, Bonin F, Becker H, Randerath WJ, Stieglitz S, Hagmeyer L, Priegnitz C, Pfeifer M, Blaas SH, Putensen C, Theuerkauf N, Quintel M, Moerer O. A novel extracorporeal CO(2) removal system: results of a pilot study of hypercapnic respiratory failure in patients with COPD. Chest. 2013 Mar;143(3):678-686. doi: 10.1378/chest.12-0228. PMID 23460154